CLINICAL TRIAL: NCT02533505
Title: A Phase 4, Randomized, Double-blind, Multicenter, Placebo-Controlled Two Way Cross-Over Study to Evaluate Changes in Oxygen Consumption and Cardiac Function in COPD Patients With Resting Hyperinflation After Administration of Symbicort pMDI 160/4.5 μg.
Brief Title: Phase IV O2 Consumption Study in COPD Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D589CC00014
Record Dates: First submitted 2015-07-30; First posted 2015-08-26 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Respiratory; COPD; O2 Consumption
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort pressurized Metered Dose Inhaler (pMDI) (Active Comparator): Symbicort pressurized Metered Dose Inhaler (pMDI)
  Interventions: Drug: Budesonide 160 mcg and formoterol fumarate dihydrate 4.5 mcg Inhalation aerosol
- Placebo of reference drug (Placebo Comparator): Placebo of reference drug
  Interventions: Drug: Matching Placebo pMDI 160/4.5 μg

INTERVENTIONS:
Drug: Budesonide 160 mcg and formoterol fumarate dihydrate 4.5 mcg Inhalation aerosol — Subjects will receive a single dose (2 inhalations) of Symbicort pMDI 160/4.5 μg (2 inhalations; total dosage 320/9.0 μg) or placebo (with a spacer) in a cross-over design (a total of 2 doses of Symbicort and 2 doses of placebo over the duration of the study), and assessments will be made before and after dosing at specified timepoints
  Arms: Symbicort pressurized Metered Dose Inhaler (pMDI)
Drug: Matching Placebo pMDI 160/4.5 μg — Placebo will be given according at the same dose and schedule as the active comparator - cross-over design.
  Arms: Placebo of reference drug

SUMMARY:
A Phase IV study evaluating changes in oxygen consumption and cardiac function in Subjects with Chronic obstructive pulmonary disease (COPD) with resting hyperinflation after administration of Symbicort pMDI 160/4.5 μg.

DETAILED DESCRIPTION:
Patients with moderate/severe COPD are known to have static hyperinflation and to develop dynamic hyperinflation during exercise. Treatment with inhaled long-acting beta agonists and combination of the long-acting beta agonist (LABA), formoterol and the inhaled corticosteroid, budesonide has been shown to improve IC and decrease lung hyperinflation. In a similar previous pilot single centre study with budesonide/formoterol (Symbicort®) the analysis of cardiac outcomes demonstrated a decrease in maximum volume of oxygen (VO2) compared to placebo. Findings suggested that the use of Symbicort can decrease the cost of breathing and therefore reduce the cardiac demand experienced by COPD patients with hyperinflation at rest. The aim of this study is to investigate whether Symbicort therapy can decrease resting VO2 by decreasing static lung hyperinflation in subjects with COPD and to evaluate changes in cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent form (ICF) prior to any study specific procedures, including withholding of medications.
2. Male or female, aged 40 to 80 years, inclusive, at Screening (Visit 1).
3. Has a clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2014 guidelines with a post bronchodilator FEV1/FVC <0.7 at Screening (Visit 1).
4. Has a post-bronchodilator FEV1 ≤65% of predicted value at Screening (Visit 1). National Health and Nutrition Examination Survey (NHANES) predicted normal standards will be used for all subjects.
5. Has an increase in IC of >10% after the administration of 1 inhalation of open-label Symbicort pMDI administered with a spacer at Screening (Visit 1).
6. Has a cigarette smoking history of more than 10 pack-years (number of cigarettes smoked per day × number of years smoked)/20).
7. Be able to understand and comply with study requirements, as judged by the Investigator.

Exclusion Criteria:

1. Subject is an employee or relative of an employee involved in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous enrollment or randomization in this study.
3. Participation in another clinical study with an investigational product (IP) during the last 30 days prior to Screening (Visit 1).
4. Subjects who are unable to discontinue their regular chronic COPD medications (including LAMAs and/or LABA/ICS) and/or who are unable or unwilling to comply with study requirements.
5. Subjects who are taking uLABAs (indacaterol, vilanterol) or uLABA-containing products.
6. Subjects who are taking PDE-4 inhibitors (roflumilast).
7. Subjects who are taking oral corticosteroids on a chronic, regular basis.
8. Subjects using daytime oxygen therapy.
9. Subjects who are currently pregnant (confirmed with positive pregnancy test) or breast feeding.
10. History of respiratory tract infection (including the upper respiratory tract) and/or pulmonary exacerbation within 6 weeks prior to Screening (Visit 1).
11. Pulmonary resection or lung volume reduction surgery within 12 months prior to Screening (Visit 1), or history of lung transplantation, or, in the Investigator's opinion, the subject may need thoracotomy or other lung surgery during the study.
12. History or current diagnosis of asthma and/or alpha 1 anti-trypsin deficiency.
13. Known active tuberculosis.
14. History of interstitial lung or massive pulmonary thromboembolic disease.
15. History of bronchiectasis secondary to respiratory diseases other than COPD (eg, cystic fibrosis, Kartagener's syndrome, etc).
16. Any clinically significant disease or disorder (eg, cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, psychiatric, major physical impairment) which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, may influence the results of the study, or may affect the subject's ability to participate in the study.
17. Recent (within 12 months prior to Screening [Visit 1]) history of myocardial infarction, recent history of heart failure (New York Heart Association [NYHA] class III and IV, pulmonary edema, and/or cardiac arrhythmia.
18. Previous or current history of lung cancer.
19. History of cancer (within 5 years prior to Visit 1), except for non-metastatic, non melanoma skin cancer.
20. Subjects who cannot perform spirometry manuevers or tolerate body plethysmography.
21. Subjects with known hypersensitivity to Symbicort, its monocomponents (budesonide or formoterol), or its excipients.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Hartford, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Spartanburg, South Carolina

REFERENCES:
- [Result] Casaburi R, Kukafka D, Cooper CB, Witek TJ Jr, Kesten S. Improvement in exercise tolerance with the combination of tiotropium and pulmonary rehabilitation in patients with COPD. Chest. 2005 Mar;127(3):809-17. doi: 10.1378/chest.127.3.809. PMID 15764761
- [Result] Casanova C, Cote C, de Torres JP, Aguirre-Jaime A, Marin JM, Pinto-Plata V, Celli BR. Inspiratory-to-total lung capacity ratio predicts mortality in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Mar 15;171(6):591-7. doi: 10.1164/rccm.200407-867OC. Epub 2004 Dec 10. PMID 15591470
- [Result] Diaz O, Villafranca C, Ghezzo H, Borzone G, Leiva A, Milic-Emili J, Lisboa C. Breathing pattern and gas exchange at peak exercise in COPD patients with and without tidal flow limitation at rest. Eur Respir J. 2001 Jun;17(6):1120-7. doi: 10.1183/09031936.01.00057801. PMID 11491153
- [Result] Di Marco F, Milic-Emili J, Boveri B, Carlucci P, Santus P, Casanova F, Cazzola M, Centanni S. Effect of inhaled bronchodilators on inspiratory capacity and dyspnoea at rest in COPD. Eur Respir J. 2003 Jan;21(1):86-94. doi: 10.1183/09031936.03.00020102. PMID 12570114
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] O'Donnell DE, Lam M, Webb KA. Measurement of symptoms, lung hyperinflation, and endurance during exercise in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1557-65. doi: 10.1164/ajrccm.158.5.9804004. PMID 9817708
- [Result] O'Donnell DE, Lam M, Webb KA. Spirometric correlates of improvement in exercise performance after anticholinergic therapy in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Aug;160(2):542-9. doi: 10.1164/ajrccm.160.2.9901038. PMID 10430726
- [Result] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531
- [Result] O'Donnell DE, D'Arsigny C, Fitzpatrick M, Webb KA. Exercise hypercapnia in advanced chronic obstructive pulmonary disease: the role of lung hyperinflation. Am J Respir Crit Care Med. 2002 Sep 1;166(5):663-8. doi: 10.1164/rccm.2201003. PMID 12204862
- [Result] Seibold H, Roth U, Lippert R, Kohler J, Wieshammer S, Henze E, Stauch M. Left heart function in chronic obstructive lung disease. Klin Wochenschr. 1986 May 2;64(9):433-41. doi: 10.1007/BF01727529. PMID 3713112
- [Result] Sexton WL, Poole DC. Effects of emphysema on diaphragm blood flow during exercise. J Appl Physiol (1985). 1998 Mar;84(3):971-9. doi: 10.1152/jappl.1998.84.3.971. PMID 9480959
- [Result] Sinderby C, Spahija J, Beck J, Kaminski D, Yan S, Comtois N, Sliwinski P. Diaphragm activation during exercise in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Jun;163(7):1637-41. doi: 10.1164/ajrccm.163.7.2007033. PMID 11401887
- [Result] Stewart RI, Lewis CM. Cardiac output during exercise in patients with COPD. Chest. 1986 Feb;89(2):199-205. doi: 10.1378/chest.89.2.199. PMID 3943379
- [Result] Synn A, Pinto-Plata V, Perham C, Celli B, Divo M. Improvement in cost of breathing after use of budesonide/formoterol in COPD patients with static hyperinflation. Presented at The American Thoracic Society International Conference, May 16-21, 2014.
- [Result] Vassaux C, Torre-Bouscoulet L, Zeineldine S, Cortopassi F, Paz-Diaz H, Celli BR, Pinto-Plata VM. Effects of hyperinflation on the oxygen pulse as a marker of cardiac performance in COPD. Eur Respir J. 2008 Nov;32(5):1275-82. doi: 10.1183/09031936.00151707. Epub 2008 Jun 11. PMID 18550609
- [Result] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Result] Yan S, Kaminski D, Sliwinski P. Reliability of inspiratory capacity for estimating end-expiratory lung volume changes during exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Jul;156(1):55-9. doi: 10.1164/ajrccm.156.1.9608113. PMID 9230726
- [Derived] Divo MJ, DePietro MR, Horton JR, Maguire CA, Celli BR. Metabolic and cardiorespiratory effects of decreasing lung hyperinflation with budesonide/formoterol in COPD: a randomized, double-crossover, placebo-controlled, multicenter trial. Respir Res. 2020 Jan 20;21(1):26. doi: 10.1186/s12931-020-1288-3. PMID 31959167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites in the United States (US) between 25 August 2015 and 12 August 2016.
Pre-assignment Details: This was a Phase 4, randomized, double-blind, multi-center, placebo-controlled, 2 way cross over study to evaluate changes in oxygen consumption and cardiac function in COPD patients with resting hyperinflation after administration of Symbicort pMDI. The study consisted of 5 site visits and 1 phone visit for a total study duration of 6 weeks.
Groups:
- Symbicort pMDI/Placebo/Symbicort pMDI/Placebo; Placebo/Symbicort pMDI/Placebo/Symbicort pMDI: The study utilized a 2-treatment, 4-period, cross-over design with 2 sequences. Each patient was randomized to 1 of 2 sequences (ABAB or BABA), where 'A', 'B' denote the active treatment or placebo treatment, respectively. Patients randomized to sequence ABAB received treatment A, B, A, and B at Visit 2 to Visit 5, respectively. Patients randomized to sequence BABA received B, A, B, and A at Visit 2 to Visit 5, respectively.
Period: Overall Study
Arm/Group | Symbicort pMDI/Placebo/Symbicort pMDI/Placebo | Placebo/Symbicort pMDI/Placebo/Symbicort pMDI
Started | 26 | 25
Completed | 23 | 24
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Over All
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (8.32) [45 to 79]
Age, Customized [Number; unit: Participants]
  <50 | 3
  >=50 - <65 | 27
  >=65 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  Black Or African American | 13
  Other | 1
  White | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Oxygen Consumption (VO2; Obtained Via a Metabolic Cart)
Description: For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: Assessment (60 minutes pre and post dose) at Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), and Visit 5 (Day 21); change from baseline pre-dose to Day 21 post-dose reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Groups:
- Symbicort pMDI; Placebo: The study utilized a 2-treatment, 4-period, cross-over design with 2 sequences. Each patient was randomized to 1 of 2 sequences (ABAB or BABA), where 'A', 'B' denote the active treatment or placebo treatment, respectively. Patients randomized to sequence ABAB received treatment A, B, A, and B at Visit 2 to Visit 5, respectively. Patients randomized to sequence BABA received B, A, B, and A at Visit 2 to Visit 5, respectively.
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
mL/min | 11.366 [5.148 to 17.584] | 1.252 [-4.867 to 7.371]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — All p-values ≤ 0.05 after rounding will be considered statistically significant; Mean Difference (Final Values) = 10.114, 95% CI 2-sided [2.943 to 17.286]

2. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Oxygen Pulse (Defined as VO2/Heart Rate [HR]; VO2 is Obtained Via a Metabolic Cart; Used as a Surrogate for Stroke Volume)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/beats/min
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
mL/min/beats/min | 0.256 [0.166 to 0.345] | 0.168 [0.081 to 0.256]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; Test type: Superiority; p = 0.111, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [-0.021 to 0.196]

3. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Gas Exchange Parameter HR
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ΔHR: beats/min
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
ΔHR: beats/min | -2.481 [-3.709 to -1.253] | -2.831 [-4.049 to -1.614]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔHR; Test type: Superiority; p = 0.609, Mixed Models Analysis; Mean Difference (Final Values) = 0.350, 95% CI 2-sided [-1.018 to 1.719]

4. Secondary Outcome: Change From Pre-dose (Visit 2)to Post-dose (Visit 5) Assessment in Spirometry.
Description: Forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and IC (using an slow vital capacity [SVC] maneuver; IC/total lung capacity [TLC] will be used as a measure of resting hyperinflation). For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: FEV1: L; ΔFVC: L; ΔIC: L
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
FEV1: L; ΔFVC: L; ΔIC: L
  ΔFEV1 | 0.187 [0.151 to 0.224] | -0.004 [-0.040 to 0.033]
  ΔFVC | 0.259 [0.196 to 0.322] | -0.052 [-0.115 to 0.011]
  ΔIC | 0.256 [0.210 to 0.302] | -0.024 [-0.070 to 0.022]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔFEV1; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.191, 95% CI 2-sided [0.150 to 0.233]
Statistical Analysis 2: Comparison: Symbicort pMDI vs Placebo; ΔFVC; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.312, 95% CI 2-sided [0.236 to 0.388]
Statistical Analysis 3: Comparison: Symbicort pMDI vs Placebo; ΔIC; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.280, 95% CI 2-sided [0.218 to 0.342]

5. Secondary Outcome: Change in Vt/Ti
Description: Change from pre-dose (Visit 2) to post-dose (Visit 5) assessment in mean inspiratory flow (tidal volume [Vt]/inspiratory time [Ti]). For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Population: Units of measure: Vt/Ti: mL/sec
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/sec
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
mL/sec | 26.533 [6.730 to 46.335] | 3.217 [-16.349 to 22.784]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔVT/Ti; Test type: Superiority; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = 23.315, 95% CI 2-sided [3.723 to 42.907]

6. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in the Modified Borg Scale for Dyspnea
Description: For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo). Modified Borg scale for dyspnea was self-administered at Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), and Visit 5 (Day 21). The Borg scale is a 1-item instrument through which a subject reports dyspnea symptoms on a scale of 0-10 to quantify the intensity of dyspnea (where 10 is most intense).
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
units on a scale | -0.452 [-0.703 to -0.202] | -0.248 [-0.499 to 0.003]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; Test type: Superiority; p = 0.106, Mixed Models Analysis; Mean Difference (Final Values) = -0.204, 95% CI 2-sided [-0.454 to 0.045]

7. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Gas Exchange Parameter VCO2
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ΔVCO2: mL/min
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
ΔVCO2: mL/min | 5.994 [-1.277 to 13.264] | -4.251 [-11.417 to 2.915]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔVCO2; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 10.245, 95% CI 2-sided [2.469 to 18.021]

8. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Gas Exchange Parameter SaO2
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: SaO2: %
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
SaO2: % | 0.422 [0.034 to 0.810] | 0.181 [-0.206 to 0.568]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔSaO2; Test type: Superiority; p = 0.333, Mixed Models Analysis; Mean Difference (Final Values) = 0.242, 95% CI 2-sided [-0.255 to 0.738]

9. Secondary Outcome: Change in RR
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ΔRR: breaths/min
Measure: Least Squares Mean (95% Confidence Interval); unit: breaths/min
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
breaths/min | -0.193 [-0.691 to 0.305] | -0.430 [-0.920 to 0.060]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔRR; Test type: Superiority; p = 0.484, Mixed Models Analysis; Mean Difference (Final Values) = 0.237, 95% CI 2-sided [-0.439 to 0.913]

10. Secondary Outcome: Change in Ti/Ttot
Description: Change from pre-dose (Visit 2) to post-dose (Visit 5) assessment in fractional inspiratory time (Ti/total cycle time [Ttot]). For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Population: ΔTi/Ttot is measured as a ratio.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
ratio | 0.012 [-0.003 to 0.027] | -0.004 [-0.019 to 0.011]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔTi/Ttot; Test type: Superiority; p = 0.113, Mixed Models Analysis; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.004 to 0.036]

11. Secondary Outcome: Change in Vt
Description: Change from pre-dose (Visit 2) to post-dose (Visit 5) assessment in tidal volume (Vt). For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Population: Units of measure: ΔVt: mL
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
mL | 71.904 [47.804 to 96.005] | 14.281 [-9.475 to 38.036]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔVt; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 57.624, 95% CI 2-sided [29.701 to 85.546]

12. Secondary Outcome: Change in Ve
Description: Change from pre-dose (Visit 2) to post-dose (Visit 5) assessment in minute ventilation (Ve). For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Population: Units of measure: ΔVe: mL/min.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
mL/min | 838.232 [449.034 to 1227.431] | -23.924 [-410.389 to 362.541]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Placebo; ΔVe; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 862.157, 95% CI 2-sided [439.817 to 1284.496]

13. Secondary Outcome: Change From Pre-dose (Visit 2) to Post-dose (Visit 5) Assessment in Spirometry.
Description: FEV1/FVC. For all outcome measures, treatment group estimates are LS Means across visits (change between 2 or more time points, calculated as the value at the later time point minus the value at the earlier time point, e.g. LS means across visits up to Visit 5 minus pre-dose Visit 2 value). Estimate for difference = LS Mean (Symbicort pMDI 160mcg/4.5ug) - LS Mean (placebo).
Time Frame: as for outcome 1
Population: ΔFEV1/FVC calculated as ratio.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Symbicort pMDI | Placebo
Number analyzed (Participants) | 51 | 51
ratio | 0.017 [0.008 to 0.026] | -0.002 [-0.011 to 0.007]
Statistical Analysis 1: Comparison: Symbicort pMDI; ΔFEV1/FVC; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 0.019, 95% CI 2-sided [0.005 to 0.033]

ADVERSE EVENTS:
Arm/Group | Symbicort pMDI | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/51
Other Adverse Events (participants affected / at risk) | 13/51 | 11/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symbicort pMDI (N=51) | Placebo (N=51)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symbicort pMDI (N=51) | Placebo (N=51)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No